CLINICAL TRIAL: NCT05637489
Title: Patient Initiated Note About Goals
Acronym: PING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00110933
Record Dates: First submitted 2022-11-21; First posted 2022-12-05 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Parallel RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Patients receive PING administered by RN
  Interventions: Behavioral: PING
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: PING — Brief survey of goals and preferences
  Arms: Treatment

SUMMARY:
This is a randomized controlled trial of the Patient-Initiated Note about Goals (PING).

DETAILED DESCRIPTION:
The PING is a brief survey designed to elicit patients' goals, preferences, and preferred surrogate decision-maker. In the PING study, patients will be assigned to receive either a nurse-administered PING or usual care. Outcomes include PING completion, subsequent goals of care conversations with providers, and healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for Annual Wellness Visit at participating clinic

Exclusion Criteria:

* Non-English speaking

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with subsequent goals of care conversation | 2 months
  Conversation documented in EHR (electronic health record)

CONTACTS AND LOCATIONS:
Overall Officials: David J Casarett, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Health, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No